CLINICAL TRIAL: NCT04716998
Title: A Controlled Study to Evaluate the Safety and Efficacy of Allogeneic MesenCure for the Treatment of Pulmonary Manifestations in Patients With COVID19
Brief Title: Safety and the Efficacy of MesenCure for the Treatment of Pulmonary Manifestations of COVID-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BonusBio Group Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CP-MCS-01
Record Dates: First submitted 2021-01-17; First posted 2021-01-20 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The treatment group consisted of 50 patients, treated with MesenCure in addition to the standard of care (SoC).
  A retrospective control group based on historical data of 150 matching subjects meeting the eligibility criteria and treated with SoC alone was included, following algorithmic stratifications against the treatment group based on gender, age, and comorbidities. The control group consisted of patients hospitalized during the same year as the treatment group and in the same medical centers as the treatment group patients. The control group patients closely resembled those in the treatment group, with similar or lower ordinal clinical scores and frequencies of comorbidities, helping to avoid bias in favor of the treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MesenCure treatment (Experimental): Clinical interventions:
  Health questionnaire, respiratory rate, heart rate, blood pressure, RA O2 saturation, x-ray.
  Blood tests: leukocyte and lymphocyte count, CRP, D-Dimer, renal and liver function, optional: cytokine levels.
  Interventions: Biological: MesenCure
- Retrospective control group (No Intervention): A retrospective control group based on historical data of 150 matching subjects meeting the eligibility criteria and treated with SOC alone was included, following algorithmic stratifications against the treatment group based on gender, age, and comorbidities. The control group consisted of patients hospitalized during the same year as the treatment group and in the same medical centers as the treatment group patients. The control group patients closely resembled those in the treatment group, with similar or lower ordinal clinical scores and frequencies of comorbidities, helping to avoid bias in favor of the treatment group.

INTERVENTIONS:
Biological: MesenCure — Three administrations of MesenCure in addition to standard care
  Arms: MesenCure treatment

SUMMARY:
An open label clinical study to evaluate the safety and the efficacy of MesenCure, an allogeneic cell therapy product, for the treatment of the pulmonary manifestations in COVID19 patients

DETAILED DESCRIPTION:
Primary endpoint: The IV administration of MesenCure is safe under the following conditions: in subjects hospitalized with COVID19 moderate to severe disease, defined upon clinical situation and radiologic findings.

Secondary endpoint: The IV administration of MesenCure is efficacious under the following conditions:

Clinical parameters: Health questionnaire, respiratory rate, heart rate, blood pressure, RA O2 saturation, hospitalization duration.

______________________________________________________ Laboratory findings: leukocyte and lymphocyte count, CRP, D-Dimer, renal and liver function, optional: cytokine levels.

______________________________________________________ Radiologic findings: pulmonary infiltrates, pleural effusion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are able and agree to sign informed consent form before any study-specific procedure.
2. Males or females, age range 18-80.
3. Female subjects are eligible only if of non-child bearing potential.
4. Documented COVID19
5. O2 Saturation of ≤93%
6. Stable hemodynamic condition (blood pressure of systolic <180mm Hg and diastolic <110mm Hg)
7. Evidence of COVID19-related pulmonary infiltrates on chest X-ray/thoracic tomography.

Exclusion Criteria:

General:

1. Pregnant or breast-feeding females.
2. History of drug abuse.
3. Heavy smokers (above 2 packages a day).
4. Subjects incapable of giving consent.

Background medical conditions:

1. Known history of any significant medical disorder, which in the investigator's judgment contraindicates the subject's participation.
2. History of significant heart diseases, renal failure (estimated GFR of <30 ml/min/1.73 m2 at screening), or hepatic disease (hepatic insufficiency classified as Child-Pugh B or C).
3. Known autoimmune diseases.
4. Received any investigational drug within 30 days prior to screening day (Visit 1) (Remdesivir is not considered investigational, and is not an exclusion criteria).
5. Immunocompromised condition from any reason, at screening.
6. Abnormal clinically significant laboratory test findings, as per the investigator's judgment.
7. Poorly controlled diabetic subjects (HbA1c > 9%).
8. Known active lung malignancy.

Concomitant treatment:

1. Currently treated with Immunosuppressive agents other than corticosteroids used for treating COVID19.
2. Treatment for cancer (i.e. chemotherapy or radiotherapy treatment) within the last 12 months.

Hypersensitivity:

1. Known history of hypersensitivity to Dextran-40 (HypoThermosol®).
2. Known history of hypersensitivity to Human Serum Albumin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Safety of Mesencure | 30 days
  No treatment-related adverse reactions

SECONDARY OUTCOMES:
Improvement in RA-O2 saturation | 14 days
  Elevation to 94% and above
Elevation of lymphocytes level | 14 days
  Elevation compared to day 0
Reduction of CRP | 14 days
  Reduction compared to day 0
Improvement of health questionnaire | 21 days
  Improvement compared to day 0
Reduced hospitalization duration | 30 days
  Reduced compared to clinical site matching historical data
improvement in pulmonary infiltrates/ pulmonary congestion | 30 days
  Improvement compared to day 0

OTHER OUTCOMES:
30-day mortality rate | 30 days
  The morality rate (%) was monitored in the treatment group and compared with the the mortality rate of retrospective control group
Progressing to invasive ventilation | The latest of: four (4) weeks or until patient release from hospital.
  The proportion of the patients progressing to invasive ventilation was measured in the treatment group and compared to the proportion of retrospective control group patient progressing to invasive ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Shadi Hamoud, MD, Principal Investigator — Rambam Health Care Campus
Locations (3):
- Israel (3):
  - Kaplan Medical Center, Rehovot, Israel
  - BARUCH PADEH Medical Center, Poriya, Tiberias, Israel
  - Rambam Health campus, Haifa

IPD SHARING:
Plan to Share IPD: No